CLINICAL TRIAL: NCT00217009
Title: A Randomized Controlled Trial of Narrowband Ultraviolet B vs Topical Psoralen Plus Ultraviolet A Photochemotherapy for Hand and Foot Dermatoses
Brief Title: Study to Compare Different Light Therapies (Narrowband Ultraviolet B vs PUVA) for Hand and Foot Skin Diseases.
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unfortunately we had unforeseen difficulty recruiting to this study. Therefore we have decided to halt the study and not publish the results.
Sponsor: Mayo Clinic (Other)
Responsible Party: Mark D Davis, M.D, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2435-04
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis; Psoriasis | interventions — Therapeutics; Ficusin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Narrowband Ultraviolet B (TL-01UVB) Therapy (Active Comparator): treatments - 3x weekly for 15 months
  Interventions: Procedure: Narrowband Ultraviolet B (TL-01UVB) Therapy
- Topical Psoralen plus ultraviolet A (PUVA) (Active Comparator): Treatments - 3x weekly for 15 months
  Interventions: Procedure: Topical Psoralen plus ultraviolet A (PUVA)

INTERVENTIONS:
Procedure: Narrowband Ultraviolet B (TL-01UVB) Therapy
  Arms: Narrowband Ultraviolet B (TL-01UVB) Therapy
Procedure: Topical Psoralen plus ultraviolet A (PUVA)
  Arms: Topical Psoralen plus ultraviolet A (PUVA)

SUMMARY:
Hand and foot skin diseases, such as dermatitis and psoriasis, that do not respond to topical creams can be treated with ultraviolet light therapy. Topical psoralen plus ultraviolet A (PUVA) is commonly used to treat these conditions, but requires additional time for the hands and feet to soak in psoralens before the light treatment. Newer narrowband ultraviolet B (NBUVB) units have become available which allow for light treatment without soaking first. The purpose of this study is to determine if NBUVB is as effective as PUVA for hand and foot skin diseases.

ELIGIBILITY:
Inclusion Criteria:

Bilateral hand or foot skin disease (dermatitis, psoriasis, etc.) with symmetric distribution and severity.

Exclusion Criteria:

Age <18 years Pregnancy Liver disease Kidney disease History of skin cancer Phototherapy or systemic therapy for the skin condition in the preceding 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of treatments required to reach clearance | Baseline to 15 months

SECONDARY OUTCOMES:
Change in symptom score (erythema, scaling/hyperkeratosis, papular/vesicular eruption, and fissures) | Baseline to 15 months
Change in global score | Baseline to 15 months
Number of patients reaching clearance | Baseline to 15 months
Adverse effects | Baseline to 15 months
Number of days in remission | Baseline to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Davis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States